CLINICAL TRIAL: NCT03043625
Title: Effect of Visceral Manipulation on Electromyographic Activity of the Upper Trapezius Muscle, Cervical Range and Pain in Patients With Non-specific Neck Pain With Functional Dyspepsia: A Randomized, Double-blinded, Sham-controlled, Study
Brief Title: Visceral Manipulation Treatment to Patients With Non-specific Neck Pain With Functional Dyspepsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Collaborators: Andréia Cristina de Oliveira Silva (Unknown); Claudia Santos Oliveira (Unknown); Daniela Aparecida Biasotto-Gonzalez (Unknown); Marco Antônio Fumagalli (Unknown); Cid André Fidelis de Paula Gomes (Unknown)
Responsible Party: Principal Investigator, Fabiano Politti, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VM-2016
Record Dates: First submitted 2017-02-01; First posted 2017-02-06 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-02

CONDITIONS: Neck Pain; Functional Dyspepsia
Keywords: Neck pain; visceral manipulation; functional dyspepsia; electromyography; pain
MeSH Terms: conditions — Neck Pain; Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: randomized, double-blinded, sham-controlled, study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visceral manipulation Group (VMG) (Experimental): The VMG wil be treated with visceral manipulation to the stomach and liver
  Interventions: Other: Visceral manipulation
- Control group (CG) (Placebo Comparator): The CG will be received placebo treatment. In the placebo treatment, the therapist should place the hands over the navel region without exerting any local tension for 1 minute.
  Interventions: Other: Control group (CG)

INTERVENTIONS:
Other: Visceral manipulation — Participants will be instructed to lie down comfortably on a stretcher in the supine position, with lower limbs flexed and abdomen exposed, and the physiotherapist positioned to the right side of the patient. The therapeutic intervention will be began with the left hand of the physiotherapist in contact with the lower region of the stomach, to which a force will be applied so that the organ was moved in an upper and lateral left direction while the right hand controlled and directed the knees of the patient to the right side until the moment when the physiotherapist notice an increase in tension in the stomach region. For the liver manipulation, the same procedures will be followed, however, with contact in the right epigastric region and the knees directed to the left side. The same position will be maintained for each organ treated until the physiotherapist could feel, through touch, a decrease in the tension of the viscera. The mean treatment time will 5 minutes.
  Arms: Visceral manipulation Group (VMG)
Other: Control group (CG) — The CG will be received placebo treatment. In the placebo treatment, the therapist should place the hands over the navel region without exerting any local tension for 1 minute.
  Arms: Control group (CG)

SUMMARY:
Background: Non-specific neck pain (NS-NP) is characterized by pain in structures located in the region between the superior nuchal line and the spinal process of the first thoracic vertebra, without association with any specific systemic disease provided by multifactorial and/or little known causes.

Objective: The objective of the present study will be to verify the clinical effects of MV through visceral nociceptive inhibition in NS-NP patients with functional dyspepsia.

Methods: In this study sixty NS-NP patients with functional dyspepsia (age: 18 and 50 years) will be randomized in into two groups: visceral manipulation group (VMG) (n =30) and control group (CG) (n =30). The VMG will be treated with visceral manipulation to the stomach and liver wile CG received placebo treatment. The immediate effects and 7 days after treatment will be evaluated through pain, cervical range, and electromyographic activity of the upper trapezius.

ELIGIBILITY:
Inclusion Criteria:

* history of neck pain for a minimal period of the three months;
* neck with restricted movement (active or passive) in at least one direction;
* Neck Disability Index considering score range of 11-24 (score out of a 50) ;
* numerical rating scale (NRS) for perceived pain intensity considering 3-7 points on an 11-point;
* Presence of symptoms related to functional dyspepsia, according to the Rome III diagnostic criteria: uncomfortable postprandial fullness, early satiety, epigastric pain and epigastric burning, accompanied by no evidence of structural disease capable of explaining the symptoms .

Exclusion Criteria:

* Individuals with history of neurological disorders (i.e., irradiated pain) or neck surgery; systemic disease; connective tissue disorder and herniated disc;
* current pregnancy;
* medical diagnosis of fibromyalgia;
* physical therapy treatment with, massage, or acupuncture in the previous two weeks;
* use of analgesic, muscle relaxant, psychotropic agent, or anti-inflammatory agent in the previous three days;
* chronic neck pain resulting from a traumatic incident; chronic musculoskeletal condition (e.g., muscular disorder, polyarthritis).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-01-30 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity assessed with Numerical Rating Scale | 12 months
  Numerical rating scale (NRS) (11 point; 0: no pain, 10: the worst possible pain imaginable) translated and cross-culturally adapted for the Brazilian population
Pain area documented on a body chart | 12 months
  Pain area will documented on a body chart. The drawings will be subsequently digitized and pain areas will be measured using open source software named ImageJ (version 1.43, National Institutes of Health, Bethesda, Maryland).

SECONDARY OUTCOMES:
Electromyography | 12 months
  The sEMG signal of the upper trapezius muscle will be recorded on the side with the greatest self-reported pain.
Cervical range of motion | 12 months
  A flexometer (Sami ®) will be used to verify cervical range of motion (ROM) of the flexion/extension, right and left lateral flexion and rotation.

IPD SHARING:
Plan to Share IPD: No
The data will not be shared with other researchers. The results of the study will be published as a manuscript in a scientific journal.

REFERENCES:
- [Background] Binder A. The diagnosis and treatment of nonspecific neck pain and whiplash. Eura Medicophys. 2007 Mar;43(1):79-89. PMID 17369782
- [Result] Barral JP, Mercier P. Visceral Manipulation. Eastland Press; 2005.